CLINICAL TRIAL: NCT00927953
Title: Phase 2, Stratified, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Safety and Efficacy of MGAWN1 in Subjects With Laboratory-documented West Nile Fever or Suspected Central Nervous System Infection Due to West Nile Virus
Brief Title: Treatment of West Nile Virus With MGAWN1
Acronym: PARADIGM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early termination due to the inability to enroll (13 of 120 subjects enrolled)
Sponsor: MacroGenics (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP-MGAWN1-02
Expanded Access: NCT01206504 (No longer available)
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Results first posted 2012-11-07 (Estimated); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: West Nile Neuroinvasive Disease; West Nile Virus Infection; Encephalitis; Meningitis; Acute Flaccid Paralysis; West Nile Fever
Keywords: West Nile virus; WNV; Encephalitis; Meningitis; Acute Flaccid Paralysis; Monoclonal Antibody; WNND; West Nile Fever; WNF
MeSH Terms: conditions — West Nile Fever; Encephalitis; Meningitis; acute flaccid myelitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MGAWN1 (Experimental): 30 mg/kg single intravenous infusion of MGAWN1
  Interventions: Biological: MGAWN1
- Placebo - Normal Saline (Placebo Comparator): single intravenous infusion of saline placebo
  Interventions: Biological: Placebo - normal saline

INTERVENTIONS:
Biological: MGAWN1 — Humanized monoclonal to West Nile virus. Dose = 30 mg/kg actual body weight intravenous, one dose at Day 0.
  Arms: MGAWN1
Biological: Placebo - normal saline — Normal Saline intravenous, volume same as active comparator, one dose at Day 0
  Arms: Placebo - Normal Saline

SUMMARY:
This study will test a drug called MGAWN1 for the treatment of West Nile infections.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the safety, efficacy, and pharmacokinetics of MGAWN1 in subjects with West Nile Fever or a syndrome compatible with West Nile Neuroinvasive Disease (WNND) [encephalitis, meningitis, or acute flaccid paralysis]. Subjects can be enrolled based on a syndrome compatible with WNND, and do not need documented West Nile virus infection.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent
2. Be >=18 years of age at the time of enrollment
3. Have West Nile Fever defined as:

   1. temperature >38°C, headache, AND
   2. positive diagnostic test for WNV Ribonucleic acid or Immunoglobulin M with serum or cerebrospinal fluid (CSF)

   OR have West Nile Neuroinvasive Disease (includes neurological signs and/or symptoms of West Nile meningitis, encephalitis, and/or acute flaccid paralysis), defined as:

   • West Nile encephalitis (must meet criteria a and b below)
   1. Encephalopathy (depressed or altered level of consciousness, lethargy, or personality change lasting 24 hours)
   2. CSF pleocytosis >=5 cells/mm^3

      AND/OR

      • West Nile meningitis (must meet criteria c and d)
   3. Clinical signs of meningeal inflammation, including nuchal rigidity, Kernig or Brudzinski sign, photophobia, or phonophobia
   4. CSF pleocytosis >=5 cells/mm^3

      AND/OR

      • Acute flaccid paralysis (must meet criteria e and f)
   5. Acute onset of limb weakness with marked progression over 48 hours
   6. Two or more of the following conditions:

      * asymmetry to weakness
      * areflexia or hyporeflexia of affected limb(s)
      * absence of pain, paresthesia, or numbness in affected limb(s)
      * CSF pleocytosis >=5 cells/mm^3
      * CSF elevated protein levels (4.5 g/L)
      * electrodiagnostic studies consistent with an anterior horn cell process
      * or abnormal increased signal in the anterior gray matter as documented by spinal cord magnetic resonance imaging
4. Have epidemiological factors consistent with West Nile Virus infection (must meet criterion a or b below):

   1. Appropriate time of year for West Nile Virus transmission in region
   2. Travel history to a region where West Nile Virus is active
5. Develop signs and/or symptoms within 14 days before study enrollment.
6. If female of childbearing potential or male and in a sexual relationship with a female of childbearing potential, agree (or have partner agree) to practice abstinence or use 2 of the following methods of contraception for 120 days (approximately 4 months) after study drug administration:

   1. Oral contraceptives, or other form of hormonal birth control including hormonal vaginal rings or transdermal patches
   2. An intrauterine device
   3. Barrier contraception (condom) with a spermicide (i.e., female subject ensures use by male partner[s])
   4. Any other equivalent method of contraception (as judged by the investigator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-05; Primary Completion 2011-02 (Actual); Study Completion 2011-05 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited over two West Nile virus seasons in 2009 and 2010 at 16 (2009) to 19 (2010) sites in the United States. One participant enrolled in 2009; 12 in 2010.
Period: Overall Study
Arm/Group | MGAWN1 | Placebo - Normal Saline
Started | 6 | 7
Completed | 4 | 6
Not Completed | 2 | 1
Not completed — Death | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MGAWN1 | Placebo - Normal Saline | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 7 | 12
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (20.84) | 38.9 (18.07) | 43.5 (19.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: The Number of West Nile Neuroinvasive Disease (WNND) Participants Who Show Improvement in the Modified Rankin Scale (MRS) (>=1 Improvement in Score)
Description: The MRS is a 7-point disability scale that assesses the degree of disability in subjects with neurological impairment. Possible scores range from 0 (perfect health) up to 5 (severe disability). The scale is as follows:
  * 0 = No symptoms at all
  * 1 = No significant disability despite symptoms;
  * 2 = Slight disability;
  * 3 = Moderate disability;
  * 4 = Moderately severe disability;
  * 5 = Severe disability; bedridden, incontinent and requiring constant nursing care and attention;
  * 6 = Dead
Time Frame: Study Day 2, 7, 14, 28, and 120
Population: All randomized participants with confirmed West Nile virus infection
Measure: Number; unit: participants
Groups:
- Placebo-Normal Saline: single intravenous infusion of saline placebo
Arm/Group | MGAWN1 | Placebo-Normal Saline
Number analyzed (Participants) | 4 | 5
participants
  Day 2 | 0 | 2
  Day 7 | 1 | 3
  Day 14 | 2 | 3
  Day 28 | 2 | 4
  Day 120 | 2 | 3

2. Primary Outcome: The Number of Participants Who Had At Least 1 Treatment-Related Adverse Event
Description: Includes adverse events considered possibly, probably, or definitely related to study drug
Time Frame: 120 days
Population: Intention to treat (ITT)
Measure: Number; unit: participants
Arm/Group | MGAWN1 | Placebo - Normal Saline
Number analyzed (Participants) | 6 | 7
participants | 0 | 3

3. Secondary Outcome: The Number of Participants With a Favorable Neurologic Outcome
Description: Favorable neurologic outcome responders are defined as subjects whose Modified Rankin Score is <=2. The MRS is a 7-point disability scale that assesses the degree of disability in subjects with neurological impairment. Possible scores range from 0 (perfect health) up to 5 (severe disability). The scale is as follows:
  * 0 = No symptoms at all
  * 1 = No significant disability despite symptoms;
  * 2 = Slight disability;
  * 3 = Moderate disability;
  * 4 = Moderately severe disability;
  * 5 = Severe disability; bedridden, incontinent and requiring constant nursing care and attention;
  * 6 = Dead.
Time Frame: Study Day 2, 7, 14, 28, and 120
Measure: Number; unit: participants
Arm/Group | MGAWN1 | Placebo - Normal Saline
Number analyzed (Participants) | 4 | 5
participants
  Day 2 | 1 | 2
  Day 7 | 2 | 2
  Day 14 | 2 | 2
  Day 28 | 2 | 3
  Day 120 | 1 | 4

4. Secondary Outcome: Mean Modified Rankin Scale Scores
Description: as for outcome 1
Time Frame: Study Day 0, 2, 7, 14, 28, and 120
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MGAWN1 | Placebo - Normal Saline
Number analyzed (Participants) | 4 | 5
units on a scale
  Baseline | 3.5 (1.29) | 3.6 (1.52)
  Day 2 | 3.5 (1.29) | 2.8 (2.22)
  Day 7 | 3.3 (1.50) | 2.8 (1.92)
  Day 14 | 2.7 (2.08) | 2.5 (1.29)
  Day 28 | 2.8 (2.75) | 1.3 (1.26)
  Day 120 | 3.8 (2.87) | 2.0 (2.45)

5. Secondary Outcome: Time to a >= 1 Point Reduction in the Modified Rankin Scale Score
Time Frame: Study Day 2, 7, 14, 28, and 120
Population: Intention to treat (ITT)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | MGAWN1 | Placebo-Normal Saline
Number analyzed (Participants) | 6 | 7
Days | 14.0 [7.0 to 127.0] | 15.0 [3.0 to 40.0]

ADVERSE EVENTS:
Arm/Group | MGAWN1 | Placebo - Normal Saline
Serious Adverse Events (participants affected / at risk) | 3/6 | 1/7
Other Adverse Events (participants affected / at risk) | 5/6 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MGAWN1 (N=6) | Placebo - Normal Saline (N=7)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Encephalitis viral (Infections and infestations) | 1 (1) | 0 (0)
Meningitis viral (Infections and infestations) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MGAWN1 (N=6) | Placebo - Normal Saline (N=7)
Activated PTT prolonged (Investigations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (3)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Blood albumin decreased (Investigations) | 0 (0) | 1 (1)
Blood bicarbonate increased (Investigations) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Convulsion (Nervous system disorders) | 1 (1) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Drug withdrawal syndrome (General disorders) | 1 (1) | 0 (0)
Haematocrit decreased (Investigations) | 0 (0) | 2 (2)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0)
Irritability (General disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Mean cell haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Protein total decreased (Investigations) | 0 (0) | 1 (1)
Prothrombin time prolonged (Investigations) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tinea versicolour (Infections and infestations) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination due to the inability to enroll (only 13 of 120 subjects enrolled); leading to small numbers of subjects analyzed and therefore many pre-specified analyses were not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days